CLINICAL TRIAL: NCT05638685
Title: The Bodily Complaints Barometer: A Survey to Investigate the Impact of the Corona Measures and of Contracting a COVID-19 Infection on the Body.
Brief Title: The Bodily Complaints Barometer: The Impact of the Corona Measures and of Contracting a COVID-19 Infection on the Body.
Acronym: COVID-MSK
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702021000576
Record Dates: First submitted 2022-03-29; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: COVID-19 infection; Lockdown measures; muskuloskeletal complaints; fatigue; observational study
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dutch-speaking people living or working in Belgium: Every participant was asked to complete a questionnaire about the impact of a COVID-19 infection and/or the impact of lockdown measures as a result of the COVID-19 pandemic on fatigue and musculoskeletal complaints.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire comprises demographics, job or school related questions, screen work questions, the International Physical Activity Questionnaire (IPAQ) and questions about the participant's health.

SUMMARY:
Since December 2019, a new corona virus (SARS-CoV-2) causing COVID-19 disease, has expeditiously spread over the entire globe. Almost a half billion people caught the disease, and in those who survived, it soon became clear that residual complaints are not rare phenomena. Early focus lay on diminished lung capacity and cardiovascular-related problems. As time passed however, it became more apparent that those are not the only residual symptoms survivors may experience.

Furthermore, nearly every country in the world took some sort of lockdown measures in order to try contain the spreading of the virus. These measures had great impact on all inhabitants, infected with the virus or not.

This questionnaire-based study therefore aims to investigate (a) the effects of a COVID-19 infection on fatigue and/or musculoskeletal complaints, new or already existing, but also (b) the effects of lockdown measures on fatigue and/or musculoskeletal complaints, new or already existing, in people living, working or studying in Belgium during the pandemic.

DETAILED DESCRIPTION:
Since the start of the COVID-19 pandemic, almost half a billion people worldwide were infected with the new coronavirus, SARS-CoV-2, causing COVID-19 disease. In Belgium, 3.6 million people, a third of the population, contracted the disease. More than 30.000 patients did not survive this condition.

Many of those who did survive, however, complained of residual symptoms, even long after their infection. Initially the most reported and investigated complaints were lung and respiratory issues, but as time progressed, it became clear these were not the only residual problems after infection. A great deal of ex-patients reported lasting fatigue and musculoskeletal complaints, both myalgia and arthralgia, after they were deemed 'cured' and therefore discharged from the hospital. Since these complaints only became apparent when patients tried to resume their daily life outside the hospital, condsiderably less attention was given to these symptoms by clinicians and researchers. Therefore, this research aims to investigate the effects of a COVID-19 infection on fatigue and/or musculoskeletal complaints, both new or already existing.

In Belgium, as in many other countries all over the world, lockdown measures were installed to contain the spread of the virus. For certain periods, this meant an obligation to work from home and moreover, to only leave home for vital reasons. Before the pandemic, "telework" was rather exceptional; in a survey from September 2019, only 22% of respondents worked from home, and for just 1 day a week. So for many employees, this meant a hard transition from a fully ergonomic work space to an unadapted home environment. For those who used to walk or bike to work, physical activity levels dropped. Even more so since all sports and recreational facilities were ordered to close. Regardless of having to live through a COVID-19 infection, all these measures were of great impact on the population, and on their levels of physical activity. A second aim of this resaerch is thus to investigate the effect of lockdown measures on fatigue and/or musculoskeletal complaints, both new or already existing, in people living, working or studying in Belgium during these measures.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Living and/or working in Belgium
* Dutch speaking

Exclusion Criteria:

* Being younger than 18 years of age
* Not working or living in Belgium during the pandemic and lockdown measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dutch-speaking people working or living in Belgium at the time of the pandemic and the lockdown measurements.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal complaints following a COVID-19 infection, through the International Physical Activities Questionnaire (IPAQ). | 3 months
Fatigue following a COVID-19 infection, through the Checklist Individual Strength (CIS). | 3 months
Musculoskeletal complaints caused by lockdown measures, through the IPAQ and the Short Inventory to Monitor Psychosocial Hazards. | 3 months
  No prior COVID-19 infection
Fatigue caused by lockdown measures, through the CIS and the Short Inventory to Monitor Psychosocial Hazards. | 3 months
  No prior COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Prof, Study Director — Ghent University, Pain in Motion
Locations (1):
- Ghent University, vakgroep revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wrzesinski,D.& Kluppels, L. (2020) Telewerken gedurende COVID-19.Hoe beleven telewerkers het al of niet gedwongen thuiswerken? Brussel, België: Vias institute -INNO_DSU_MOBI
- See also: Sciensano — https://www.sciensano.be/nl/gezondheidsonderwerpen/coronavirus
- See also: World Health Organisation — https://covid19.who.int/